CLINICAL TRIAL: NCT01276743
Title: Study of Protein Tyrosine Phosphatase Non-receptor Type 22 (PTPN22) C1858T Polymorphism in Children and Adolescents of Greek Origin With Type 1 Diabetes Mellitus (T1DM)
Brief Title: Study of PTPN22 C1858T Polymorphism in Children and Adolescents of Greek Origin With T1DM
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Styliani Giza, MD, MSc, PhD, 4th Department of Pediatrics, Faculty of Medicine, Aristotle University of Thessaloniki, Papageorgiou General Hospital, Thessaloniki, Greece, Aristotle University Of Thessaloniki
Other Study IDs: 01051979
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- T1DM: Children and adolescents with T1DM
- Unaffected Population: Population not known to be affected by T1DM

SUMMARY:
The protein tyrosine phosphatase non-receptor type 22 (PTPN22) gene encodes a lymphoid-specific phosphatase (LYP) which is an important downregulatory factor of T cell activation. A PTPN22 polymorphism, C1858T, was found associated with T1DM in different Caucasian populations.

In this observational case-control study, we aimed at confirming the role of PTPN22, C1858T polymorphism in T1DM predisposition in a Greek population.

ELIGIBILITY:
Inclusion Criteria:

For the patients

* Diagnosis of T1DM according to American Diabetes Association (ADA) Criteria as well as according to International Society for Pediatric and Adolescent Diabetes (ISPAD) Guidelines
* Unrelated male and female subjects
* 1-20 years of age
* Come from Greece (At least 3 grandparents are Greek)
* At least one year post onset of T1DM
* Sign written informed consent

Inclusion Criteria:

For the controls

* Unrelated nondiabetic male and female subjects with no family history of T1DM
* Equal to or greater than 18 years of age
* Come from Greece (At least 3 grandparents are Greek)
* Be screened by a questionnaire to ensure the absence of any diagnostic evidence of autoimmune diseases or family history (first- or second-degree relatives) of T1DM
* Sign written informed consent

Exclusion Criteria:

For the patients •Subjects who do not meet the criteria above

Exclusion Criteria:

For the controls

•Subjects who do not meet the criteria above

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents of Greek origin who attended the Pediatric Diabetes Outpatient Clinic of 4th Department of Pediatrics of Medical School of Aristotle University of Thessaloniki for T1DM
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
• Difference of distribution of PTPN22 C1858T alleles between patients and controls of Greek origin | 3 years

SECONDARY OUTCOMES:
• The association between PTPN22 C1858T polymorphism among patients and gender | 3 years
• The association between PTPN22 C1858T polymorphism among patients and age of onset of type 1 diabetes mellitus (T1DM) | 3 years
• The association between the PTPN22 C1858T polymorphism among patients and presence of autoantibodies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, MD, PhD, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism, 4th Department of Pediatrics, Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece